CLINICAL TRIAL: NCT05350618
Title: Developing Novel Ultrasound Techniques for Assessing the Pelvic Myofascial Tissues to Investigate Their Involvement in Provoked Vestibulodynia
Brief Title: Pelvic Floor Myofascia: A New Player Involved in Vulvodynia
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Full Professor, Université de Sherbrooke
Other Study IDs: MP-31-2021-4165
Record Dates: First submitted 2022-04-07; First posted 2022-04-28 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy; Vulvodynia
Keywords: Fascia; Pelvic floor; Provoked vestibulodynia; Pain; Sexual dysfunctions; Ultrasound
MeSH Terms: conditions — Vulvodynia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic controls: A single transperineal ultrasound assessment session will be conducted by two independent physiotherapists with an expertise in pelvic floor rehabilitation
  Interventions: Other: Ultrasound evaluation
- Women with provoked vestibulodynia: A single transperineal ultrasound assessment session will be conducted by one physiotherapist with an expertise in pelvic floor rehabilitation
  Interventions: Other: Ultrasound evaluation

INTERVENTIONS:
Other: Ultrasound evaluation — A single transperineal ultrasound assessment session

SUMMARY:
This study aims to develop novel ultrasound evaluation techniques to characterize the different pelvic myofascial tissues and to examine the intra- and inter-rater reliability of these techniques (objective 1). Moreover, the potential contribution of the pelvic myofascial tissues to the etiology of provoked vestibulodynia will be investigated by comparing the ultrasound data of women with provoked vestibulodynia to that of asymptomatic controls (objective 2). Women interested in participating in the study will contact the research assistant for a screening interview over the phone. Eligible women will then be invited to take part in a pelvic floor ultrasound assessment session at the Urogynecology Research Laboratory. For the first objective, asymptomatic controls will be evaluated by two independent physiotherapists with an expertise in pelvic floor rehabilitation. Intra- and inter-rater reliability of ultrasound data will be analyzed. For the second objective, asymptomatic controls and women with a diagnosis of provoked vestibulodynia will be evaluated by an expert physiotherapist specialized in pelvic floor rehabilitation. Differences in ultrasound data between the two groups will be analyzed.

DETAILED DESCRIPTION:
Vulvodynia, chronic vulvar pain, is identified as a neglected condition by the World Health Organization and the National Institutes of Health. This is explained by a poor understanding of the pathology and compromised diagnosis, leading to poor therapeutic management and a lack of effective treatment options. Provoked vestibulodynia, characterized by pain at the entry of the vagina elicited by pressure and penetration, is the leading subtype of vulvodynia. Recent scientific advances have highlighted the importance of the pelvic floor muscles and the potential role of the surrounding connective tissues (the fascias). Therefore, a new potential contributor is emerging in the etiology of provoked vestibulodynia, namely the pelvic myofascial tissues. The first objective of this study is to develop transperineal ultrasound evaluation techniques (B-mode and ultrasound elastography/shearwave) to assess the morphometry (thickness) and viscoelasticity (shear strain and shear elastic modulus) of the pelvic myofascial tissues and to examine the intra- and inter-rater reliability in asymptomatic controls. The second objective of this study is to examine the potential contribution of the pelvic myofascial tissues to the etiology of provoked vestibulodynia. To do this, morphometric (thickness) and viscoelastic (shear strain and shear elastic modulus) ultrasound imaging features of the pelvic myofascial structures will be compared in women with provoked vestibulodynia and asymptomatic controls. The association between ultrasound data and clinical characteristics will also be investigated. The clinical characteristics will include self-administered psychosexual questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* No pain during sexual intercourse (for the healthy women)
* Moderate to severe pain (≥ 5/10) during sexual intercourse for at least 3 months (for women with provoked vestibulodynia)
* Moderate to severe pain (≥ 5/10) at least 90% of the time when engaging in or attempting sexual intercourse for at least 3 months (for women with provoked vestibulodynia)

Exclusion Criteria:

* Current or past pregnancy
* Urogynecological condition (e.g., pelvic organ prolapse stage ≥ 3, urinary leakage, current urinary/vaginal infection or in the last 3 months)
* Other causes of vulvo-vaginal pain (e.g., spontaneous vulvovaginal pain not related to sexual intercourse/contact, dermatological condition, herpes, vulvo-vaginal atrophy)
* Post-menopausal state
* Previous vulvar, vaginal or pelvic surgery (e.g., vestibulectomy, pelvic organ prolapse surgery)
* Physiotherapy within the last 9 months
* More than 3 physiotherapy treatment within last year
* Medication that could influence pain perception (e.g., analgesic, antidepressant)
* Other medical conditions that could interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic controls (without any vulvar pain) and women suffering from provoked vestibylodynia (moderate to severe pain for at least 90% of the time when engaging in or attempting sexual intercourse) are being recruited.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Morphometry - muscle thickness | Baseline evaluation
  Muscle thickness will be measured by transperineal ultrasound in B-mode.
Viscoelasticity - shear strain | Baseline evaluation
  Shear strain will be measured by transperineal ultrasound with elastography.
Viscoelasticity - shear elastic modulus | Baseline evaluation
  Shear elastic modulus be measured by transperineal ultrasound with elastography/shearwave.

SECONDARY OUTCOMES:
Pain intensity | Baseline evaluation
  To assess pain intensity during intercourse (Numerical Rating Scale (NRS), ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain possible).
Pain quality | Baseline evaluation
  To assess pain quality including its sensory, affective and evaluative components using the McGill-Melzack pain questionnaire (MPQ). Minimum value: 0, Maximum value: 78, higher scores indicate worse pain.
Depression symptoms | Baseline evaluation
  To address depressive symptoms according to the Beck Depression Inventory (BDI-II). Minimum value: 0, Maximum value: 63, higher scores indicate more severe depression symptoms.
Sexual function | Baseline evaluation
  To assess sexual function using the Female Sexual Function Index (FSFI). Minimum value: 2, Maximum value: 36, Inferior scores indicate lower sexual function.
Sexual distress | Baseline evaluation
  To assess sexual distress (Female Sexual Distress Scale - FSDS). Minimum value: 0, Maximum value: 52, Superior scores indicate higher sexually related distress.
Pain catastrophizing | Baseline evaluation
  Pain catastrophizing assessed with the Pain Catastrophizing Scale (PCS). Minimum value: 0, Maximum value: 52, Superior scores indicate higher pain catastrophizing.
Fear of pain | Baseline evaluation
  Fear of pain according to the Pain Anxiety Symptoms Scale (PASS-20). Minimum value: 0, Maximum value: 100, Superior scores indicate higher fear of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided